CLINICAL TRIAL: NCT05717153
Title: Intratumoral Extracellular Metabolic Impact of DFMO and AMXT 1501
Brief Title: Intratumoral Extracellular Metabolic Impact of DFMO and AMXT 1501 in Patients With Diffuse or High Grade Glioma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 22-005690; NCI-2022-10375 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R37CA276851 (NIH)
Record Dates: First submitted 2023-01-23; First posted 2023-02-08 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Diffuse Glioma; Malignant Glioma
MeSH Terms: conditions — Glioma | interventions — Specimen Handling; Eflornithine; Magnetic Resonance Spectroscopy; Microdialysis; Drug Implants

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The patient and the principal investigator will be blinded to each patient's assignment until after the catheter has been placed. However, the clinical research coordinators and co-investigators will remain unblinded to facilitate study coordination and ensure protocol adherence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Arm I (MRI, resection, DFMO, AMXT 1501) (Experimental): Patients undergo magnetic resonance imaging (MRI) and surgical resection at baseline. Patients receive eflornithine PO in combination with AMXT 1501 PO on days 1-5 post-surgery. Patients also undergo CT after surgery and collection of blood on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Eflornithine; Procedure: Magnetic Resonance Imaging; Drug: Polyamine Transport Inhibitor AMXT-1501 Dicaprate; Procedure: Resection; Device: Microdialysis; Procedure: Placement
- Arm II (MRI, resection, placebo, DMFO, AMXT 1501) (Placebo Comparator): Patients undergo magnetic MRI and surgical resection at baseline. Patients receive placebo PO on days 1 and 2 post-surgery, and then receive eflornithine PO and AMXT 1501 PO on days 3-5 post-surgery. Patients also undergo CT after surgery and collection of blood on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Eflornithine; Procedure: Magnetic Resonance Imaging; Drug: Polyamine Transport Inhibitor AMXT-1501 Dicaprate; Procedure: Resection; Device: Microdialysis; Procedure: Placement
- Arm III (MRI, resection, DMFO, AMXT 1501) (Active Comparator): Patients undergo magnetic MRI and surgical resection at baseline. Patients receive eflornithine PO alone on days 1 and 2 post-surgery, then receive eflornithine PO in combination with AMXT 1501 PO on days 3-5 post-surgery. Patients also undergo CT after surgery and collection of blood on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Eflornithine; Procedure: Magnetic Resonance Imaging; Drug: Polyamine Transport Inhibitor AMXT-1501 Dicaprate; Procedure: Resection; Device: Microdialysis; Procedure: Placement

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Eflornithine — Given PO
  Other Names: Alpha-Difluoromethylornithine; DFMO; Difluoromethylornithine; Difluromethylornithine
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Drug: Polyamine Transport Inhibitor AMXT-1501 Dicaprate — Given PO
  Other Names: AMX 513 Dicaprate; AMX513 Dicaprate; AMXT 1501 Dicaprate; AMXT-1501 Dicaprate
Procedure: Resection — Undergo surgical resection
  Other Names: Surgical Resection
Device: Microdialysis — Undergo Microdialysis
Procedure: Placement — Undergo placement of catheters
  Other Names: Place

SUMMARY:
This early phase I trial studies brain tumor (glioma) metabolism in response to eflornithine (DFMO) and polyamine transport inhibitor AMXT-1501 dicaprate (AMXT 1501) in patients with diffused or high grade glioma. Brain tumors use and produce certain molecules to survive and grow. DFMO is an irreversible inhibitor of ornithine decarboxylase, the enzyme catalyzing polyamine synthesis. AMXT 1501 is a polyamine transport inhibitor which prevents uptake of polyamines from the extracellular environment. This trial is being done to analyze how DFMO and AMXT 1501 affect brain tumor metabolism based on the molecules in the tumor's fluid.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine how polyamine depletion impacts extracellular guanidinoacetate abundance.

SECONDARY OBJECTIVES:

I. Determine the impact of polyamine depletion on polyamine abundance and the global extracellular metabolome within live human gliomas, in situ.

II. Assess the feasibility of longitudinal microdialysis to evaluate pharmacodynamic responses of in situ gliomas to therapeutic intervention in a post-operative setting.

III. Assess the central nervous system (CNS) pharmacokinetics of DFMO and AMXT 1501.

IV. Adverse effects of study drugs in the immediate postoperative setting during microdialysis.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients undergo surgical resection with magnetic resonance imaging (MRI) and placement of catheters for microdialysis at baseline. Patients receive DFMO orally (PO) in combination with AMXT 1501 PO on days 1-5 post-surgery in the absence of disease progression or unacceptable toxicity. Patients also continue microdialysate collection as well as undergo computed tomography (CT) and collection of blood on study.

ARM II: Patients undergo surgical resection with MRI and placement of catheters for microdialysis at baseline. Patients receive DFMO PO and AMXT 1501 PO on days 3-5 post-surgery in the absence of disease progression or unacceptable toxicity. Patients also continue microdialysate collection, as well as undergo CT and collection of blood on study.

ARM III: Patients undergo surgical resection with MRI and placement of catheters for microdialysis at baseline. Patients receive DFMO PO alone on days 1 and 2 post-surgery, then receive eflornithine PO in combination with AMXT 1501 PO on days 3-5 post-surgery in the absence of disease progression or unacceptable toxicity. Patients also continue microdialysate collection, as well as undergo CT and collection of blood on study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Clinical and radiographic evidence suggesting a diagnosis of a diffuse high grade glioma (HGG), or a prior diagnosis of a diffuse glioma
* Planned subtotal resection or biopsy due to tumor location, size, or other clinical indication deemed appropriate by the surgeon
* Provide written informed consent for the current study and the Neuro-Oncology biorepository for archiving of cerebrospinal fluid (CSF) and blood samples collected on this protocol. Willing to remain in the hospital at Mayo Clinic (Rochester, MN) for three days added to their standard post-operative stay to undergo longitudinal microdialysis
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L without transfusion within 7 days preceding the lab assessment (obtained =< 14 days prior to registration)
* Platelet >= 100 x 10^9/L, without transfusion within 7 days preceding the lab assessment (obtained =< 14 days prior to registration)
* Hemoglobin >= 9 g/dL, without transfusion support within 7 days preceding the lab assessment (obtained =< 14 days prior to registration)
* Activated partial thromboplastin time or partial thromboplastin time (aPTT or PTT) =< 1.5 x upper limit of normal (ULN) (obtained =< 14 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN (obtained =< 14 days prior to registration)
* Total serum bilirubin =< 1.5 x ULN (obtained =< 14 days prior to registration)
* The patient is clinically euthyroid [Thyroid Stimulating Hormone (TSH)]
* Serum creatinine =< 1.5 x ULN or creatinine clearance >= 60 mL/min/1.73 m^2 for patients with serum creatinine levels above 1.5 x ULN (obtained =< 14 days prior to registration)
* Negative serum or urine pregnancy test is required for female subjects of childbearing age < 14 days prior to registration

Exclusion Criteria:

* Inappropriate surgical candidates due to current or past medical history or uncontrolled concurrent illness which limits safety of or compliance to study proceedings
* Vulnerable populations: pregnant or nursing women, prisoners, mentally handicapped
* Unable to swallow tablets or who are at risk for impaired absorption of oral medication. NOTE: This includes but not limited to, refractory vomiting, gastric resection/bypass, and duodenal/jejunal resection
* Known hypersensitivity or allergy to DFMO or AMXT 1501
* Contraindication to MRI or administration of gadolinium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in the tumor/brain extracellular guanidinoacetate ratio | Baseline up to 2 months
  Targeted metabolomics will be performed using the microdialysate aliquot collected at each time point to quantify guanidinoacetate content. Fold change values will be calculated between each time point within a patient. Fold changes values between time points will be compared across the three arms for statistically significant differences using a Wilcoxon signed rank test; p < 0.05 will be considered statistically significant.

SECONDARY OUTCOMES:
Measured extracellular levels of glutamate in tumor and brain microdialysates | Up to 2 months
  Targeted metabolomics will be performed for each time point's microdialysate, assaying for polyamines (putrescine, spermine, and spermidine), in addition to ornithine and glutamate. Fold change values will be calculated between each time point within a patient. Fold changes values between time points will be compared across the three arms for statistically significant differences using a Wilcoxon signed rank test; p < 0.05 will be considered statistically significant.
Proportion of longitudinal microdialysis aliquots containing > 30 uL of microdialysate | Up to post-operative day 5
  Targeted metabolomics will be performed for each time point's microdialysate, assaying for polyamines (putrescine, spermine, and spermidine), in addition to ornithine and glutamate. Fold change values will be calculated between each time point within a patient. Fold changes values between time points will be compared across the three arms for statistically significant differences using a Wilcoxon signed rank test; p < 0.05 will be considered statistically significant.
Central nervous system free drug levels from microdialysate - DFMO | Up to 2 months
  Drug levels of difluoromethylornithine (eflornithine [DFMO]) at each time point will be calculated for pharmacokinetic analyses by Aminex Therapeutics to determine time of peak concentration (hr), maximum drug concentration (ng/mL), and area under the curve 0-t (hr*ng/mL).
Central nervous system free drug levels from microdialysate - AMXT 1501 | Up to 2 months
  Polyamine transport inhibitor AMXT-1501 dicaprate (AMXT 1501) at each time point will be calculated for pharmacokinetic analyses by Aminex Therapeutics to determine time of peak concentration (hr), maximum drug concentration (ng/mL), and area under the curve 0-t (hr*ng/mL).
AMXT 1501 brain/plasma ratio over time | Up to 2 months
  Will be assessed via longitudinal microdialysis to understand how AMXT 1501 is distributed in Central Nervous System (CNS) tissue with and without tumor as compared to plasma levels over time.
Incidence of adverse events | Up to 2 months
  Although no significant additional risks are anticipated in the proposed context, safety data will be assessed to evaluate for any unanticipated adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Terence C. Burns, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials